CLINICAL TRIAL: NCT03458624
Title: Observational Study to Evaluate the Safety and Efficacy of FURESTEM-AD Inj. in Moderate to Severe Atopic Dermatitis Patients Who Participated in Phase 1/2a Clinical Trial of FURESTEM-AD Lnj.
Brief Title: Long-term Observational Study to Evalution the Safety and Efficacy of FURESTEM-AD Inj.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Kang Stem Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: KSTHD_FURESTEM_AD_EXT
Record Dates: First submitted 2017-04-03; First posted 2018-03-08 (Actual); Last update posted 2018-03-08 (Actual); Status verified 2018-02

CONDITIONS: Atopic Dermatitis
Keywords: FURESTEM-AD Inj.; Stem cells
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Not applicable-observational study: Not applicable-observational study

SUMMARY:
Observational Study to Assess the Safety and Efficacy of FURESTEM-AD lnj. In moderate to Atopic Dermatitis

DETAILED DESCRIPTION:
This is a observational study, single center, open label, study of safety and Efficacy of FURESTEM-AD Inj. in subjects with moderate to severe Atopic Dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects participating in this observational study originally participated in study FURESTEM-RA Inj.[NCT02221258]
* Subject who understands and voluntarily sign an informed consent form

Exclusion Criteria:

* In case follow-up is not possible from end of clinical trial Phase 1/2a to end of this study period

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects participating in this observational study originally participated in study FURESTEM-AD Inj. [NCT01927705]
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2016-08-12 (Actual); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate the number of adverse events Safety of FURESTEM-AD Inj. | 3 years
  The severity of each adverse enent was classified according to CTCAE v4.0

SECONDARY OUTCOMES:
Percentage of patients who decreased more than 50% in SCORAD(SCORing of Atopic Dermatitis) INDEX compared to Phase 2a clinical trial baseline | 3 years
Variation of SCORAD Total Score as contrasted with Phase 2a clinical trial baseline value or Phase 2a clinical trial closing value | 3 years
Percentage of subjects whose IGA(Investigator's Global Assessment) evaluation results were reduced to zero or one point | 3 years
Variation of serum Total IgE as contrasted with Phase 2a clinical trial baseline value or Phase 2a clinical trial closing value | 3 years
Variation of EASI(Eczema area and severity index) as contrasted with Phase 2a clinical trial baseline value or Phase 2a clinical trial closing value | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Tae-Yun Kim, Principal Investigator — Seoul St. Mary's Hospital
Locations (1):
- Seoul ST. Mary's Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No